CLINICAL TRIAL: NCT04360642
Title: Singing for Wellness: Is Singing a Useful Way of Supporting People in South Devon to Self-manage Aspects of Their COPD: Does a Bespoke Respiratory Choir Provide a Non-medical Intervention for Those With COPD in Our Local Community
Brief Title: Singing for Wellness: Is Singing a Useful Way of Supporting People in South Devon to Self-manage Aspects of Their COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 209103
Record Dates: First submitted 2019-01-25; First posted 2020-04-24 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Singing

STUDY DESIGN:
Intervention Model Description: Singing for Wellness will use an uncontrolled observational study design. Two mixed-cohort, 12-week community choirs will be delivered by experienced vocal practitioners in South Devon localities: Newton Abbott and Torquay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- singing arm (Other): Singing for Wellness will use an uncontrolled observational study design. Two mixed-cohort, 12-week community choirs will be delivered by experienced vocal practitioners in South Devon localities: Newton Abbott and Torquay.
  Lung function, frailty and health-related quality of life will be assessed by Spirometry, CRQ (chronic respiratory questionnaire), MRC breathlessness scale, Rockwood frailty and Warwick-Edinburgh Mental Well-being Scale (WEMWBS). Participants will be assessed at baseline and then again at completion of the 12-week course.
  Written feedback from participants to capture qualitative experience using narrative and Patient Reported Outcome Measures (PROMs). The attrition and attendance rate will also be recorded for later review.
  Interventions: Other: singing

INTERVENTIONS:
Other: singing — Singing for Wellness will use an uncontrolled observational study design. Two mixed-cohort, 12-week community choirs will be delivered by experienced vocal practitioners in South Devon localities:

SUMMARY:
The aim of this study is to explore whether singing is a useful way of supporting people in South Devon to self manage aspects of their COPD and associated social isolation. It will also investigate whether a model of bespoke respiratory community choirs provides a useful service for our local community. The study will look at the impact of singing on breathing, wellbeing, frailty and engagement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD

  * Evidence of airflow obstruction as measured by spirometry
  * Being independently mobile and able to get to location
  * Being able to give permission to participate
  * Over 18 years old
  * Awaiting pulmonary rehabilitation or have completed pulmonary rehabilitation

Exclusion Criteria:

* Lacking capacity to give permission to participate e.g. severe dementia

  * Other health issues which preclude participation e.g. psychosis, unstable physical health
  * Under 18 years of age
  * Not diagnosed with COPD

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Lung function | 12 weeks
  Lung function will be assessed by Spirometry (FVC and FEV1)
Lung function | 12 weeks
  Lung function will be assessed by Medical Research Council (MRC) breathlessness scale (Scores 1-5, good to worse)
Lung function | 12 weeks
  Lung function will be assessed by Chronic Respiratory Questionnaire (CRQ), Likert scale 1-7, higher scores indicate better health related quality of life

SECONDARY OUTCOMES:
Mental Wellbeing | 12 weeks
  Warwick-Edinburgh Mental Wellbeing Scale which assesses the mental wellbeing (positive mental health) of a person.(scores 1-5 experiences from none of the time to all of the time)
Frailty | 12 weeks
  Rockwood Frailty Scale to categories a patient into one of nine general frailty classifications.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Roberts, Study Director — Torbay and South Devon NHS Foundation Trust
Locations (1):
- Torbay Hospital, Torquay, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No